CLINICAL TRIAL: NCT06566456
Title: The Impact of Modified Site for Radial Artery Cannulation on the Stability of Arterial Blood Pressure Monitoring
Brief Title: Effect of Modified Radial Artery Cannulation Site on IABP Monitoring Stability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025ZSLYEC-505
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-01

CONDITIONS: Perioperative Arterial Pressure Monitoring
Keywords: Radial Artery Cannulation, Modified Cannulation Site ，Catheter Stability, Invasive Blood Pressure Monitoring, arterial catheter function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.5-2.5 cm proximal to the radial styloid process (Experimental): The ultrasound-guided radial artery puncture site is1.5-2.5 cm proximal to the radial styloid process
  Interventions: Procedure: The puncture site is 1.5-2.5 cm proximal to the radial styloid process
- traditional site (Active Comparator): The ultrasound-guided radial artery puncture site is level with the radial styloid process and where the radial artery pulse is most prominent
  Interventions: Procedure: traditional site

INTERVENTIONS:
Procedure: The puncture site is 1.5-2.5 cm proximal to the radial styloid process — The ultrasound-guided radial artery puncture site is1.5-2.5 cm proximal to the radial styloid process
  Arms: 1.5-2.5 cm proximal to the radial styloid process
Procedure: traditional site — The ultrasound-guided radial artery puncture site is level with the radial styloid process and where the radial artery pulse is most prominent
  Arms: traditional site

SUMMARY:
Invasive arterial blood pressure (IABP) monitoring is critical for perioperative and critically ill patients, yet traditional radial artery cannulation near the wrist joint is prone to catheter dysfunction (e.g., kinking, occlusion) due to positional changes, compromising accuracy and patient safety. This trial hypothesizes that modifying the cannulation site to 1.5-2.5 cm proximal to the radial styloid process may enhance catheter stability.

DETAILED DESCRIPTION:
Methods and analysis:This is a prospective, parallel-group, randomized, controlled, analyst-blinded trial. A total of 486 participants (231 per group, adjusted for 5% dropout) will be enrolled. Eligible patients (18-75 years, ASA physical status I-III, requiring elective surgery with radial artery cannulation) will be randomized 1:1 to the modified group (1.5-2.5 cm proximal to the radial styloid process) or the conventional group (traditional site). The primary outcome is the incidence of arterial catheter dysfunction (defined by criteria such as blood sampling difficulty, position-dependent waveform, or improved waveform post-square wave test). Secondary outcomes include frequency of catheter dysfunction, damping abnormality rate, first-puncture success rate, number of arterial punctures,arterial cannulation time, complication incidence, and blood pressure measurement differences.

Sample size calculation:This trial utilized a superiority test for sample size calculation. In the 100-case preliminary experiment results, the incidence rate of abnormal arterial catheter function was 30% in the control group and 12% in the modified group. With a predefined superiority margin Δ of -6% (actual observed Δ of -18%), using a type I error rate (α) of 0.025 and statistical power (1-β) of 0.90, statistical calculations determined that 231 participants per group (totaling 462) would be required to detect this difference in a two-sided test. Considering a 5% dropout rate among study subjects, the final planned sample size was adjusted to 486 cases.

ELIGIBILITY:
Inclusion criteria

1. Patients 18-75 years of age undergoing elective surgery who require radial artery cannulation;
2. Patients positioned in supine, lithotomy, or other face-up surgical postures;
3. American Society of Anesthesiologists (ASA) physical status classification: Grades I to III.

Exclusion criteria

1. Abnormal results from the modified Allen test;
2. Patients with a history of radial artery cannulation within the past 3 months, or with infection/trauma at or adjacent to the puncture site;
3. Coagulopathy or hypercoagulable state;
4. Patients undergoing anticoagulant therapy;
5. Comorbid vascular diseases (e.g., vasculitis);
6. Patients undergoing surgical procedures involving the same anatomic region;
7. Preoperative hemodynamic instability (including patients already on vasoactive medications, or with atrial fibrillation, atrial flutter, atrioventricular block of grade II or higher, multifocal ventricular premature beats, or ventricular premature beats with R-on-T phenomenon);
8. Patients lacking legal capacity to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of arterial catheter dysfunction | during the period of catheter indwelling
  (a) difficulty in blood sampling: When drawing arterial blood samples for blood gas analysis, the sample cannot be aspirated smoothly through the arterial pressure monitoring line, necessitating repeated flushing of the line to obtain an adequate sample; or arterial catheter occlusion occurs and a new arterial pressure monitoring pathway must be established based on surgical or anesthetic requirements; (b) position-dependent waveform or flushing: repositioning of the arterial catheter or wrist is required to obtain a satisfactory arterial waveform, or smooth flushing can only be achieved following such repositioning. (c) improved waveform post-square wave test: after a square wave test (conducted every 30 minutes or when the arterial waveform becomes flat), the arterial waveform shows significant improvement compared to its pre-flush state.

SECONDARY OUTCOMES:
Frequency of arterial catheter dysfunction | during the period of catheter indwelling
  mean number of catheter instability events per subject per hour.
Damping abnormality rate and frequency | during the period of catheter indwelling
  Damping abnormality rate: the ratio of total cases with over-damping or under-damping to the total number of enrolled patients per group.
  Damping abnormality frequency: mean number of over-damping or under-damping events per subject per hour.
First-puncture success rate | From the start of arterial puncture until successful arterial catheter placement or abandonment of the arterial catheter placement procedure,up to 10 minutes
  the ratio of cases with successful first-time arterial cannulation to the number of enrolled cases per group. A successful first puncture is defined as achieving arterial access and catheter placement without needle withdrawal or repositioning after initial skin entry.
Number of arterial punctures | From the start of arterial puncture until successful arterial catheter placement or abandonment of the arterial catheter placement procedure,up to 10 minutes
  total number of arterial punctures performed before successful cannulation. One puncture is defined as withdrawing the needle to the subcutaneous layer and reinserting it during the cannulation process.
Arterial Cannulation Time | From the start of arterial puncture until successful arterial catheter placement or abandonment of the arterial catheter placement procedure,up to 10 minutes
  defined as the interval from the first skin entry of the needle to the first display of an arterial blood pressure waveform on the monitor.
Complication incidence | from the time of the puncture onset until the time of every day after arterial puncture (at 1-day, 2-day, 3-day
  encompasses complications during puncture and catheter indwelling (e.g., hematoma, bleeding, ecchymosis) and post-puncture complications (e.g., bleeding, hematoma, distal ischemia, local infection, peripheral nerve injury, unintended catheter dislodgment). The observation window is 0-3 days post-surgery.
Difference in IABP before and after square wave test. | during the period of catheter indwelling
  The difference between the invasive blood pressure value before wave test and the invasive blood pressure value after waveform stabilization
Difference between IABP and NIBP | during the period of catheter indwelling
  The difference between the invasive blood pressure value and the cuff pressure after waveform stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Sanqing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (2):
- China (2):
  - the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews FJ, Nolan JP. Critical care in the emergency department: monitoring the critically ill patient. Emerg Med J. 2006 Jul;23(7):561-4. doi: 10.1136/emj.2005.029926. PMID 16794104
- [Background] Chatterjee A, DePriest K, Blair R, Bowton D, Chin R. Results of a survey of blood pressure monitoring by intensivists in critically ill patients: a preliminary study. Crit Care Med. 2010 Dec;38(12):2335-8. doi: 10.1097/CCM.0b013e3181fa057f. PMID 20890190
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Araghi A, Bander JJ, Guzman JA. Arterial blood pressure monitoring in overweight critically ill patients: invasive or noninvasive? Crit Care. 2006;10(2):R64. doi: 10.1186/cc4896. PMID 16630359
- [Background] Antonelli M, Levy M, Andrews PJ, Chastre J, Hudson LD, Manthous C, Meduri GU, Moreno RP, Putensen C, Stewart T, Torres A. Hemodynamic monitoring in shock and implications for management. International Consensus Conference, Paris, France, 27-28 April 2006. Intensive Care Med. 2007 Apr;33(4):575-90. doi: 10.1007/s00134-007-0531-4. PMID 17285286
- [Background] Cockings JG, Webb RK, Klepper ID, Currie M, Morgan C. The Australian Incident Monitoring Study. Blood pressure monitoring--applications and limitations: an analysis of 2000 incident reports. Anaesth Intensive Care. 1993 Oct;21(5):565-9. doi: 10.1177/0310057X9302100512. PMID 8273876
- [Background] Hager HH, Burns B. Artery Cannulation(Archived). 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482242/ PMID 29489243
- [Background] Clark VL, Kruse JA. Arterial catheterization. Crit Care Clin. 1992 Oct;8(4):687-97. PMID 1327430
- [Background] Nuttall G, Burckhardt J, Hadley A, Kane S, Kor D, Marienau MS, Schroeder DR, Handlogten K, Wilson G, Oliver WC. Surgical and Patient Risk Factors for Severe Arterial Line Complications in Adults. Anesthesiology. 2016 Mar;124(3):590-7. doi: 10.1097/ALN.0000000000000967. PMID 26640979
- [Background] White L, Halpin A, Turner M, Wallace L. Ultrasound-guided radial artery cannulation in adult and paediatric populations: a systematic review and meta-analysis. Br J Anaesth. 2016 May;116(5):610-7. doi: 10.1093/bja/aew097. PMID 27106964
- [Background] Robertson-Malt S, Malt GN, Farquhar V, Greer W. Heparin versus normal saline for patency of arterial lines. Cochrane Database Syst Rev. 2014 May 13;2014(5):CD007364. doi: 10.1002/14651858.CD007364.pub2. PMID 24825673
- [Background] Alves M, Barbier C, Fangio P, Hayon J, Loubieres Y, Pichereau C, Maury E, Outin H. Arterial catheters' dysfunction according to insertion site: an observational study. Minerva Anestesiol. 2017 Feb;83(2):222-224. doi: 10.23736/S0375-9393.16.11606-2. Epub 2016 Oct 4. No abstract available. PMID 27701374
- [Background] Imbriaco G, Monesi A, Giugni A, Cilloni N. Radial artery cannulation in intensive care unit patients: Does distance from wrist joint increase catheter durability and functionality? J Vasc Access. 2021 Jul;22(4):561-567. doi: 10.1177/1129729820953020. Epub 2020 Aug 27. PMID 32854566
- [Background] Z.-N. Z ,X. L,J. L, et al.Abstract PR028: A Survey of the Incidence and Consequences of Invasive Blood Pressure Measuring Errors Caused By Arterial Line Occlusion[J].Anesthesia Analgesia,2016,123(3S2):45-45.